CLINICAL TRIAL: NCT00330421
Title: A Phase II Clinical and Correlative Study of BAY 43-9006 (Sorafenib) IND 69,896 in Sarcoma
Brief Title: Sorafenib in Treating Patients With Soft Tissue Sarcomas (Extremity Sarcoma Closed to Entry as of 5/30/07)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03122; 05-033; U01CA062490 (NIH)
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2013-11

CONDITIONS: Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Osteosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Osteosarcoma; Stage I Adult Soft Tissue Sarcoma; Stage II Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Sarcoma | interventions — Sorafenib

ARMS (2):
- Group I (sarcomas of extremity, closed accrual as of 5/30/07) (Experimental): Patients receive oral sorafenib twice daily on days 1-14. Patients undergo surgical resection of the tumor on approximately day 15. Once patients recover from surgery (and radiotherapy if indicated), patients who demonstrate a clinically and pathologically significant response (≥ 25% reduction in tumor size or ≥ 25% necrosis in the surgical specimen) may continue sorafenib as above for a maximum of 6 months in the absence of disease progression or unacceptable toxicity and at the discretion of the principal investigator. Biopsy tissue and blood samples are examined for biomarkers and interstitial fluid pressure (IFP) is measured at baseline and immediately before surgery.
  Interventions: Drug: sorafenib tosylate; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: computed tomography; Procedure: dynamic contrast-enhanced magnetic resonance imaging
- Group II (metastatic or inoperable sarcomas) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for 2 courses. Patients with responding or stable disease may continue sorafenib in the absence of disease progression or unacceptable toxicity. Biopsy tissue and blood samples are examined for biomarkers and IFP is measured at baseline and on days 28 and 56.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: computed tomography; Procedure: dynamic contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Procedure: therapeutic conventional surgery — Undergo surgery
  Arms: Group I (sarcomas of extremity, closed accrual as of 5/30/07)
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: computed tomography — Correlative studies
  Other Names: tomography, computed
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Correlative studies
  Other Names: DCE-MRI

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with soft tissue sarcoma. Sorafenib may stop the growth of soft tissue sarcoma by blocking blood flow to the tumor and blocking some of the enzymes needed for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the combined vascular endothelial growth factor receptor 2 (VEGF-R2)/platelet-derived growth factor receptor (PDGFR)-beta inhibitor BAY 43-9006/ sorafenib can decrease interstitial fluid pressure (IFP) in soft tissue sarcomas.

II. To investigate the effects of BAY 43-9006/sorafenib on tumor blood flow, circulating endothelial cells, vascular density and pericyte coverage.

III. To characterize the pharmacokinetics of BAY 43-9006/sorafenib in sarcoma patients.

SECONDARY OBJECTIVES:

I. To describe any preliminary evidence of anti-tumor activity. II. Assess whether there are any significant relationships between systemic drug exposure and drug-related toxicity or biological effect.

OUTLINE: This is a multicenter study. Patients are assigned to one of two groups (group 1 closed to accrual as of 5/30/07).

GROUP I (SARCOMAS OF THE EXTREMITY) (CLOSED TO ACCRUAL AS OF 5/30/07): Patients receive oral sorafenib twice daily on days 1-14. Patients undergo surgical resection of the tumor on approximately day 15. Once patients recover from surgery (and radiotherapy if indicated), patients who demonstrate a clinically and pathologically significant response (≥ 25% reduction in tumor size or ≥ 25% necrosis in the surgical specimen) may continue sorafenib as above for a maximum of 6 months in the absence of disease progression or unacceptable toxicity and at the discretion of the principal investigator. Biopsy tissue and blood samples are examined for biomarkers and interstitial fluid pressure (IFP) is measured at baseline and immediately before surgery.

GROUP II (METASTATIC OR INOPERABLE SARCOMAS): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for 2 courses. Patients with responding or stable disease may continue sorafenib in the absence of disease progression or unacceptable toxicity. Biopsy tissue and blood samples are examined for biomarkers and IFP is measured at baseline and on days 28 and 56.

In both groups, blood samples are drawn periodically for pharmacological studies.

After completion of study therapy, patients are followed monthly until all study-related toxicities are resolved and then at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* There are two groups of patients eligible for this study; treatment group 1 consists of patients with extremity sarcomas other than potentially curable osteosarcoma or Ewing's sarcoma who are candidates for potentially curative surgery; treatment group 2 consists of patients with metastatic or inoperable sarcoma, for which there is no known curative or survival prolonging palliative therapy, or failure of these therapies; patients must have at least one site of measurable disease by radiologic imaging techniques; patients must have at least one palpable tumor mass with no overlying viscera which is amenable to biopsy; the tumor mass should be approximately 2 cm or greater in diameter; patients with smaller palpable tumors are eligible if participation is approved by the treating surgeon after discussion with the study chairperson

  * As of 5/30/07, no subjects will accrue to Treatment Group I
* Life expectancy >= 2 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Pretreatment laboratory data, obtained within 14 days of study entry, must meet the following criteria:
* Absolute Neutrophil Count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5-times the upper limit of normal (ULN)
* Serum glutamic-pyruvic transaminase (SGPT)=< 2.5-times ULN
* Total Bilirubin =< ULN
* Serum creatinine =< 1.5-times ULN
* >= 3 weeks since major surgery unrelated to study disease (sarcoma)
* >= 3 weeks since chemotherapy or radiation therapy (6 weeks for nitrosourea or mitomycin C chemotherapy)
* No prior treatment with sorafenib (BAY 43-9006) or specific inhibitors of mitogen-activated protein kinase (MAPK) pathways are permitted; a previously irradiated tumor site cannot be used for clinical or correlative measurements, although irradiation to sites other than a measurable site is permitted; there are no limitations on the extent or type of prior therapy received by the patient other than the time intervals indicated in the above and demonstrating complete recovery from any adverse effects associated by satisfying all relevant eligibility criteria
* Patients who are on warfarin anticoagulation are allowed to participate as long as they are converted to a low molecular weight heparin (e.g. lovenox) from study entry until at least day 56
* Women of childbearing potential must not be pregnant or lactating; all women of childbearing potential (age < 50, last menstrual period [LMP] < 12 months ago) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L of beta-HCG) within 72 hr prior to receiving the study medication; BAY43-9006 has antiproliferative effects, which may be harmful to the developing fetus or nursing infant
* Fertile males and females must use adequate contraception
* Signed informed consent

Exclusion Criteria:

* Ewing's sarcoma or osteosarcoma that is potentially curable with surgery, chemotherapy, and/or radiation therapy
* Active brain metastases including evidence of cerebral edema by CT scan or MRI, or progression from prior imaging study, any requirements for steroids, or enzyme-inducing anti-convulsant agents, or clinical symptoms of/from brain metastases; patients with treated and/or stable brain metastasis who are asymptomatic can be enrolled, if otherwise eligible
* Any uncontrolled serious medical or psychiatric illness; particular note is given to uncontrolled hypertension (discretion left to investigators) and significant proteinuria > 1 gm/24 hr (does not require quantitation in absence of clinical indication)
* Patients receiving other investigational agents
* Human immunodeficiency virus (HIV) patients receiving combination anti-retroviral therapy are excluded because of potential pharmacokinetic interactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Morgan, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Raut CP, Boucher Y, Duda DG, Morgan JA, Quek R, Ancukiewicz M, Lahdenranta J, Eder JP, Demetri GD, Jain RK. Effects of sorafenib on intra-tumoral interstitial fluid pressure and circulating biomarkers in patients with refractory sarcomas (NCI protocol 6948). PLoS One. 2012;7(2):e26331. doi: 10.1371/journal.pone.0026331. Epub 2012 Feb 7. PMID 22347360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase II study enrolled pts with metastatic or inoperable sarcomas. Additional eligibility criteria: at least one site of measurable disease, at least one superficial palpable tumor (>1cm) amenable to biopsy, age ≥18 years, Eastern Cooperative Oncology Group (ECOG) performance status ≤2, and no prior sorafenib therapy.
Pre-assignment Details: Additional eligibility criteria included: at least one site of measurable disease by radiologic imaging, at least one superficial palpable tumor (>1cm) with no overlying viscera amenable to biopsy, age ≥18 years, Eastern Cooperative Oncology Group (ECOG) performance status ≤2, and no prior sorafenib therapy.
Groups:
- Group II (Metastatic or Inoperable Sarcomas): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days for 2 courses. Patients with responding or stable disease may continue sorafenib in the absence of disease progression or unacceptable toxicity. Biopsy tissue and blood samples are examined for biomarkers and IFP is measured at baseline and on days 28 and 56.
  laboratory biomarker analysis : Correlative studies
  sorafenib tosylate : Given PO
  pharmacological study : Correlative studies
  computed tomography : Correlative studies
  dynamic contrast-enhanced magnetic resonance imaging : Correlative studies
- Group I (Sarcomas of Extremity): Patients receive oral sorafenib twice daily on days 1-14. Patients undergo surgical resection of the tumor on approximately day 15. Once patients recover from surgery (and radiotherapy if indicated), patients who demonstrate a clinically and pathologically significant response (≥ 25% reduction in tumor size or ≥ 25% necrosis in the surgical specimen) may continue sorafenib as above for a maximum of 6 months in the absence of disease progression or unacceptable toxicity and at the discretion of the principal investigator. Biopsy tissue and blood samples are examined for biomarkers and interstitial fluid pressure (IFP) is measured at baseline and immediately before surgery.
Period: Overall Study
Arm/Group | Group II (Metastatic or Inoperable Sarcomas) | Group I (Sarcomas of Extremity)
Started | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group II (Metastatic or Inoperable Sarcomas)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Fludeoxyglucose (FDG) Uptake (Maximal Standardized Uptake Value, or SUVmax)
Description: Paired comparison made using a Wilcoxon signed rank test with one-sided type I error of 5%.
Time Frame: Baseline to up to 1 month post-treatment
Reporting Status: Not Posted

2. Primary Outcome: Change in Interstitial Fluid Pressure (IFP)
Description: Paired comparison made using a Wilcoxon signed rank test with one-sided type I error of 5%.
Time Frame: Baseline to up to 1 month post-treatment
Population: IFP measurements were obtained in only 6 of 15 patients at baseline. Only 2 of these 6 patients had SD at 28 and 56 days and therefore, second IFP measurements were only obtained in those 2 patients.
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Group II (Metastatic or Inoperable Sarcomas)
Number analyzed (Participants) | 2
mm Hg | 4.25 [3.0 to 5.5]

3. Primary Outcome: Change in White Blood Cell Count (WBC)
Description: Paired comparison made using a Wilcoxon signed rank test with one-sided type I error of 5%.
Time Frame: Baseline to up to 1 month post-treatment
Reporting Status: Not Posted

4. Primary Outcome: Change in Pericyte Coverage of Endothelial Cells (Alpha-SMA)
Description: Paired comparison made using a Wilcoxon signed rank test with one-sided type I error of 5%.
Time Frame: Baseline to up to 1 month post-treatment
Reporting Status: Not Posted

5. Primary Outcome: Clinical Benefit as Measured by 50% Reduction in IFP
Time Frame: Baseline to surgery
Reporting Status: Not Posted

6. Primary Outcome: Clinical Benefit, Measured by Any Reduction in Tumor Dimensions on CT Scan as Measured by RECIST Criteria
Time Frame: Up to 1 month
Reporting Status: Not Posted

7. Primary Outcome: Incidence of Adverse Events
Time Frame: Up to 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group II (Metastatic or Inoperable Sarcomas)
Serious Adverse Events (participants affected / at risk) | 11/15
Other Adverse Events (participants affected / at risk) | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group II (Metastatic or Inoperable Sarcomas) (N=15)
Fatigue (General disorders) | 11 (22) — Fatigue
Hemoglobin (Blood and lymphatic system disorders) | 8 (16) — Low hemoglobin
Alkaline phosphatase (Hepatobiliary disorders) | 7 (16) — Elevated alk phos
AST (Hepatobiliary disorders) | 7 (16) — Elevated AST
Hematologic - other (Blood and lymphatic system disorders) | 6 (11) — Other hematologic issue, including thrombocytopenia and clotting dysfunction
Diarrhea (Gastrointestinal disorders) | 6 (11) — Diarrhea without prior colostomy
Abdominal pain (Gastrointestinal disorders) | 5 (11) — Abdominal pain
Anorexia (General disorders) | 5 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group II (Metastatic or Inoperable Sarcomas) (N=15)
Hand-foot reaction (General disorders) | 7 (21) — Hand-foot reaction

LIMITATIONS AND CAVEATS:
No Grade 4 toxicities were noted (15 patients). IFP measurements were obtained in only 6 of 15 patients at baseline. Only 2 of these 6 patients had SD at 28 and 56 days and therefore, second IFP measurements were only obtained in those 2 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less